CLINICAL TRIAL: NCT03508544
Title: Evaluation of Postoperative Analgesic Effect of Ultrasound Guided Erector Spinae Plane Block and Transmuscular Quadratus Lumborum Block in Hip and Proximal Femur Surgery, Randomised Controlled Study
Brief Title: Lumbar Erector Spinae Plane Block and Quadratus Lumborum Block in Hip and Proximal Femur Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maltepe University (Other)
Responsible Party: Principal Investigator, Asst. Prof. Serkan Tulgar, M.D., Assistant Professor, Maltepe University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Lumbar ESP vs QLB
Record Dates: First submitted 2018-04-16; First posted 2018-04-25 (Actual); Last update posted 2018-06-07 (Actual); Status verified 2018-06

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lumbar ESP block (Active Comparator): Ultrasound-guided lumbar Erector spinae plane (ESP) block performed at the begining of the surgery with 40 ml of a bupivacaine/lidocaine mixture. Perioperative and postoperative routine analgesic protocol will be performed (consist of intravenous analgesics and intravenous patient-controlled analgesia) with no additional intervention (block) Standard Pain Followup and Monitorization will be performed
  Interventions: Procedure: Lumbar ESP block; Other: Standard Pain Followup and Monitorization
- QLB Block (Active Comparator): Ultrasound-guided transmuscular quadratus lumborum block (QLB) performed at the begining of the surgery with 40 ml of a bupivacaine/lidocaine mixture. Perioperative and postoperative routine analgesic protocol will be performed (consist of intravenous analgesics and intravenous patient-controlled analgesia) with no additional intervention (block) Standard Pain Followup and Monitorization will be performed
  Interventions: Procedure: QLB bLock; Other: Standard Pain Followup and Monitorization
- Control (Sham Comparator): Perioperative and postoperative routine analgesic protocol will be performed (consist of intravenous analgesics and intravenous patient-controlled analgesia) with no additional intervention (block) Standard Pain Followup and Monitorization will be performed.
  Interventions: Other: Standard Pain Followup and Monitorization

INTERVENTIONS:
Procedure: Lumbar ESP block — Lumbar ESP block will be performed at the begining of surgery under ganeral anesthesia. A convex ultrasound transducer will be placed in a longitudinal parasagittal orientation 4-6 cm lateral to L4 spinous process. The erector spinae muscles will be identified superficial to the tip of L4 transverse process. The patient's skin will be anesthetized with 2% lidocaine. A 22-gauge 10-cm needle will be inserted using an out-plane superior-to-inferior approach to place the tip into the fascial plane on the deep (anterior) aspect of erector spinae muscle. The location of the needle tip will be confirmed by visible fluid spread lifting erector spinae muscle off the bony shadow of the transverse process. A total of 40 mL of bupivacaine/lidocaine mixture will be injected.
  Arms: Lumbar ESP block
Procedure: QLB bLock — QLB block will be performed at the begining of surgery under ganeral anesthesia. The convex transducer will be placed in the transverse plane on the flank of the patient cranial to the iliac crest.The 4th lumbar vertebral transverse process, erector spinae muscles, psoas muscles, transverse abdominis muscles, internal and external oblique muscles and the quadratus lumborum muscles will be identified. A 15cm 22G insulated needle will be inserted on the posterior corner of the convex probe. 40 ml of local anesthetic mixture(bupivacaine and lidocaine ) will be administered between the quadratus lumborum and psoas muscles into the fascial plane. We observed the local anesthetic pressing down on the psoas muscle in the ultrasound image.
  Arms: QLB Block
Other: Standard Pain Followup and Monitorization — Numeric Rating Scale (NRS) pain score will be recorded from 20th minute in recovery room followed by 1.-3.-6.-12.-18.-24.hours. Intravenous meperidine administration at 0.5 mg / kg rescue analgesia was determined in patients with a NSR score of 6 and over in the postoperative collection room. It is planned that the patient will continue to follow the hourly NRS score in ward. Intramuscular diclofenac will be administered in this period if NRS 6 and if it is over, intravenous 0.5 mg / kg meperidine will be administered if NRS score is 6 or more after 2 hours. Salvage analgesic needs and times will be noted in detail, and the use of rescue analgesics, as well as NRS scores at designated hours, will be kept in a statistical evaluation.

SUMMARY:
Multimodal analgesia is used to control postoperative pain in hip surgery. Quadratus lumborum block is an effective regional anesthesia technique for hip and proximal femur surgery. The erector spinae plane block applied to the lumbar region was also reported to provide effective analgesia in these surgeons. In this study, we aimed to determine and compare the effects of quadratus lumborum block and lumbar erector spinae plane block on postoperative pain in hip and proximal femur surgeons.

ELIGIBILITY:
Inclusion Criteria:

- Hip joint and proxiaml femur surgery, ASA 1-2-3

Exclusion Criteria:

* Patient refusal
* Contraindications to regional anesthesia
* Known allergy to local anesthetics
* Bleeding diathesis
* Use of any anti-coagulants
* Inability to provide informed consent
* Severe kidney or liver disease
* Inability to operate PCA system
* Patient with psychiatric disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-04-09 (Actual); Primary Completion 2018-05-21 (Actual); Study Completion 2018-06-06 (Actual)

PRIMARY OUTCOMES:
Pain | 24 hours
  Changes in Numeric Rating Scale (NRS) at rest and on movement will be recorded at intervals. NRS is a unidimensional measure of pain intensity in adults. The NRS is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain. The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").

SECONDARY OUTCOMES:
analgesic consumption | 24 hours
  Tramadol consumption in Patient Controlled Analgesia device and additional and rescue analgesic using

CONTACTS AND LOCATIONS:
Overall Officials: Serkan Tulgar, Ass Prof, Principal Investigator — Maltepe University Faculity of Medicine
Locations (1):
- Maltepe University faculty of medicine, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tulgar S, Selvi O, Senturk O, Ermis MN, Cubuk R, Ozer Z. Clinical experiences of ultrasound-guided lumbar erector spinae plane block for hip joint and proximal femur surgeries. J Clin Anesth. 2018 Jun;47:5-6. doi: 10.1016/j.jclinane.2018.02.014. Epub 2018 Mar 6. No abstract available. PMID 29522966
- [Background] He J, Zheng XQ, Luo CH, Huang ZX, He WY, Wang HB, Yang CX. [Effects and safety of quadratus lumborum block in analgesia after hip arthroplasty]. Zhonghua Yi Xue Za Zhi. 2018 Feb 27;98(8):565-569. doi: 10.3760/cma.j.issn.0376-2491.2018.08.002. Chinese. PMID 29534382
- [Background] Ueshima H, Yoshiyama S, Otake H. RETRACTED: The ultrasound-guided continuous transmuscular quadratus lumborum block is an effective analgesia for total hip arthroplasty. J Clin Anesth. 2016 Jun;31:35. doi: 10.1016/j.jclinane.2015.12.033. Epub 2016 Mar 22. PMID 27185672 (Retraction: PMID 35393191 J Clin Anesth. 2022 Aug;79:110702; PMID 35397960 J Clin Anesth. 2022 Aug;79:110704)